CLINICAL TRIAL: NCT02711696
Title: Randomized Clincal Trial on the Effect of a Restricted Gluten Contamination Elimination Diet in Achieving Complete Mucosal Healing Among Celiac Patients With Persisting Minimal Duodenal Lesions During Gluten Free Diet [GluCED]
Brief Title: Randomized Clincal Trial on the Effect of a Restricted Gluten Contamination Elimination Diet Among Celiacs [GluCED]
Acronym: GluCED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Alberto Lanzini, MD PhD, Associate Professor of Gastroenterology, PhD, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD_GE_2013
Record Dates: First submitted 2016-03-07; First posted 2016-03-17 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Celiac Disease
Keywords: Celiac Disease,; Gluten Free Diet; Gluten contamination
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A, GCED cohort (Active Comparator): GCED, Gluten Contamination Elimination Diet
  Interventions: Behavioral: GCED, Gluten Contamination Elimination Diet
- B, time cohort (No Intervention): Cohort B consisted of patients on long term follow-up that accepted a repeated biopsies 60 or more months later the first control biopsy.

INTERVENTIONS:
Behavioral: GCED, Gluten Contamination Elimination Diet — A Gluten Free diet based exclusively on naturally gluten-free products and foods, with the elimination from the diet of all commercially available processed food and products labeled "gluten free " (Gluten Contamination Elimination Diet, GCED).
  Arms: A, GCED cohort

SUMMARY:
The study assessed whether compete healing of duodenal mucosa in celiac patients with persistent Marsh I-II lesion after 1 year of gluten free diet (GFD):

* could be achieved by adoption of a diet based exclusively on naturally gluten free products, with the elimination of commercially available processed food (GCED, Gluten Contamination Elimination Diet);
* may depend upon time of exposure to GFD.

Investigators studied two cohorts of celiac patients, both on GFD, for at least one year:

* cohort A: patients re-biopsied after three months on GCED;
* cohort B: patients re-biopsied after a minimum of further two years on standard GFD.

DETAILED DESCRIPTION:
Despite strict adherence to gluten free diet (GFD), the complete healing of the duodenal mucosa of celiac patients is rarely achieved. The cause of the persistence of the inflammation is not yet understood.

It is well known that there is a high degree of variability in individual response to gluten with some patients worsening of duodenal histology upon exposure to very small amount of gluten.

This observation suggest that contamination with gluten of commercially available processed food and/or small amount of gluten in processed foods labeled "gluten-free" (less than 20 ppm) may prevent complete mucosal healing.

This explanation is indirectly supported by a study of Hollon et al. (2013) showing that persistence of gastrointestinal symptoms in celiac patients on a GFD is abolished, in 85% of cases, by the adoption of a diet based exclusively on naturally gluten-free products, and on the elimination from the diet of commercially available processed food and products labeled "gluten free " (Gluten Contamination Elimination Diet, GCED).

The main aim of this study was to assess whether the complete healing of duodenal mucosa in patients with persistent Mars I-II lesions after 1 year on GFD i) could be achieved, as a proof of the concept, by the adoption of a GCED OR ii) may depend upon time of exposure to GFD. To achieve this aim investigators studied 2 cohorts of patients with Marsh I-II lesion after 1 year on GFD: cohort A re-byopsied after 3 month GCED , and cohort B re-biopsied after a minimum of further 2 years on standard GFD.

ELIGIBILITY:
Inclusion Criteria:

* Marsh I-II lesion at 12-18 months after starting GFD
* Negative Celiac Disease serology
* Strict adherence to gluten free diet without digression

Exclusion Criteria:

* presence of Gastrointestinal Symtoms
* presence of Helicobacter pylori infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Histologic classification | three months in cohort A, at least sixty months in cohort B
  Assessment of Marsh class (0-I-II-III) on duodenal biopsies in participants from both cohorts

SECONDARY OUTCOMES:
Celiac disease serology | three months in cohort A, at least sixty months in cohort B
  IgA t-TG (class A Antibodies anti tissue Transglutaminases) were measured in particiapnts serum at the same time of dudenal biopsy [Eu t-Tg Eurospital, Trieste, Italy]
TCR+ T cells count | three months in cohort A, sixty months in cohort B
  TCR+ T cells were identified using a commercially available method suitable for formalin fixed paraffin embedded dudenal biopsies. A mean of the count of TCR+T cells was obtained with a cut-off value of 4 out of 100 epithelial cells.
Eosinophils count | three months in cohort A, sixty months in cohort B
  Eosinophils were identified and counted on duodenal biopsies with a cut off value of 2 out of 100 epithelial cells.

CONTACTS AND LOCATIONS:
Overall Officials: barbara zanini, MD, PhD, Study Director — Università degli Studi di Brescia

IPD SHARING:
Plan to Share IPD: No